CLINICAL TRIAL: NCT01983111
Title: A Multicenter, Phase IV, Interventional Study to Compare the Efficacy and Safety of NORSPAN to Tramadol/Acetaminophen in Patients With Prolonged Postoperative Pain After Spinal Surgery (PASSION)
Brief Title: Compare the Efficacy and Safety of Norspan to Tramadol/Acetaminophen With Prolonged Postoperative Pain (PASSION)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Korea Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUP13-KR-401
Record Dates: First submitted 2013-10-14; First posted 2013-11-13 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Buprenorphine; Ultracet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- buprenorphine (Experimental): Patch
  Interventions: Drug: buprenorphine
- tramadol/acetaminophen (Active Comparator): Oral tablet
  Interventions: Drug: tramadol/acetaminophen

INTERVENTIONS:
Drug: buprenorphine — Dosage and administration: This one patch should be attached every 7 days.
  Other Names: Norspan patch
  Arms: buprenorphine
Drug: tramadol/acetaminophen — Amount of drug ingredients
  : Acetaminophen 325 mg and Tramadol hydrochloride 37.5 mg in 1 tablet of this drug.
  Dosage and administration:
  Adjust dose depending on a patient's pain severity and treatment response. Starting at the initial dose of 2 tablets, usually administer 4 tablets per dose, twice daily. At a dosing interval of at least 12 hr, the daily dose should not exceed 8 tablets.
  Other Names: Ultracet ER semi
  Arms: tramadol/acetaminophen

SUMMARY:
The purpose of this study is to compare the efficacy and safety of buprenorphine transdermal system to tramadol/acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Korean men and women aged 20 years or more
* Presence of pain associated with a spinal disease and lumbar fusion at 1-2 spinal segments (1-2 level lumbar fusion surgery)
* Moderate to severe pain of the NRS pain score ≥ 4 at Visit 1 (14~90 days after surgery, Baseline) (Amended 21Nov2013)
* Consent to participate in the study and voluntary signature on the informed consent form

Exclusion Criteria:

* Women of childbearing potential, except for the following cases:
* A partner who is vasectomized or otherwise surgically sterile.
* Use of 2 contraception methods. Two methods include the combination of double-barrier contraception or barrier contraception and hormone contraception, and appropriate barrier methods are as follows: Diaphragm (female contraceptive device), condom, intrauterine (copper or hormone), sponge or spermicide. Hormonal contraceptives include all commercially available products containing estrogen and/or progesterone.
* Pregnant or breastfeeding women. Pregnant woman is defined as a woman after fertilization to late pregnancy with a positive result from the urine pregnancy test.
* History of hypersensitivity to buprenorphine, tramadol, APAP or excipients, and celecoxib
* Medical history of asthma, acute rhinitis, nasal polyp, vascular edema urticaria or allergic reaction to aspirin or other non-steroidal anti-inflammatory drugs(NSAIDs, COX-2)
* Hypersensitivity or intolerance to Domperidone
* Risk of gastrointestinal irritation such as gastrointestinal bleeding, mechanical ileus or perforation
* Genetic problem such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Severely impaired respiratory function or respiratory depression
* Current use of monoamine oxidase(MAO) inhibitors or the medication history within 2 weeks prior to study participation
* Convulsive disorder, head injury, shock, decreased level of consciousness of uncertain origin, intracranial lesion or increased intracranial pressure or severe hepatic impairment
* Biliary tract disorder
* Presence or suspected drug abuse history
* Medical history of opioid or drug dependence
* Current use of other CNS inhibitors or muscle relaxants that may result in dyspnea, hypotension, severe sedation or coma when used with the investigational product, opioid analgesics
* Use of strong opioids, buprenorphine or tramadol/APAP within 1 week prior to study participation (however, study participation is allowed for PRN prescription of PCA and strong opioids)
* Any condition representing a contraindication of application of buprenorphine, tramadol/APAP or celecoxib
* Major pain not attributable to a spinal disease
* Anticancer therapy that may affect pain assessment
* Clinically significant cardiovascular or renal dysfunction
* Postoperative complications
* Symptoms of acute pain after lumbar fusion or characteristic analgesic features showing rapidly changing needs for analgesics
* Current use of other investigational product at enrollment or within 30 days after administration of other investigational product

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhyok Kim, Dr.PhD, Principal Investigator — Sanggye Paik Hospital, Dept. of Orthopedic Surgery
Locations (1):
- Sanggye Paik Hospital, Dept. of Orthopedic Surgery, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Kim JH, Kim JH, Kim HS, Min WK, Park YS, Lee KY, Lee JH. Efficacy and Safety of Transdermal Buprenorphine versus Oral Tramadol/Acetaminophen in Patients with Persistent Postoperative Pain after Spinal Surgery. Pain Res Manag. 2017;2017:2071494. doi: 10.1155/2017/2071494. Epub 2017 Sep 13. PMID 29056859

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol/Acetaminophen: Oral tablet
  tramadol/acetaminophen: Amount of drug ingredients
  : Acetaminophen 325 mg and Tramadol hydrochloride 37.5 mg in 1 tablet of this drug.
  Dosage and administration:
  Adjust dose depending on a patient's pain severity and treatment response. Starting at the initial dose of 2 tablets, usually administer 4 tablets per dose, twice daily. At a dosing interval of at least 12 hr, the daily dose should not exceed 8 tablets.
Period: Overall Study
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Started | 70 | 66
Completed | 58 | 59
Not Completed | 12 | 7
Not completed — Withdrawal by Subject | 8 | 6
Not completed — Adverse Event | 4 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: * Safety set = 134
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Tramadol/Acetaminophen | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 38 | 64
  >=65 years | 43 | 27 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.42 (10.84) | 61.54 (8.96) | 63.02 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 29 | 73
  Male | 25 | 36 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in the Pain Intensity Score (0-10 NRS) From Visit 1 (Baseline) to 6weeks After Treatment.
Description: NRS-Pain scale assessed the severity of a subject's pain of mean pain over the past 24 hours prior to the visit on a scale of 0 (No pain) and 10 (Worst possible pain). Change = mean score at Week6/ET minus mean score at Baseline.
Time Frame: baseline and 6 weeks
Population: In the PP set, the change in the pain intensity score from Visit 1 (Baseline) to Week 6 of the investigational product administration was analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Number analyzed (Participants) | 47 | 40
Scores on a scale | -2.32 (1.96) | -2.75 (1.56)
Statistical Analysis 1: Comparison: Buprenorphine vs Tramadol/Acetaminophen; In the Per protocol set; Test type: Non-Inferiority or Equivalence — In the PP set, for a non-inferiority test of the reduction in the pain intensity score from Visit 1 (Baseline) to Week 6 of treatment, the lower limit of the 97.5% onesided confidence interval was compared to a clinical non-inferiority margin, -1.5; p = 0.2658, t-test, 2 sided; Mean Difference (Final Values) = -0.43, 97.5% CI 2-sided [-6 to 3], Standard Deviation 1.79

2. Secondary Outcome: Change in the Pain Intensity Score (0-10 NRS) From Visit 1 (Baseline) to Week 2 of the Investigational Product Administration
Description: NRS-Pain scale assessed the severity of a subject's pain of mean pain over the past 24 hours prior to the visit on a scale of 0 (No pain) and 10 (Worst possible pain). Change = mean score at Week 2/ET minus mean score at Baseline.
Time Frame: 2 weeks
Population: In the PP set, the reduction in the pain intensity score from Visit 1 (Baseline) to Week 2 of the investigational product administration was analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Number analyzed (Participants) | 47 | 40
Scores on a scale | -1.19 (1.61) | -1.70 (1.73)

3. Secondary Outcome: Change in the Quality of Life (EQ-5D) Score From Visit 1 (Baseline) to Week 6 Post-dose
Description: EQ-5D to measure of health related quality of life should be answered as one of 3 levels about current condition for 5 dimensions for 'Motor capability', 'Self-care', 'Daily activities', 'Pain/discomfort', 'Depression/anxiety' and was calculated total average by giving a weighting on 3 level of answers (EQ-5D levels into 'no problems' (level 1) and 'problems' (level 2 and 3)).
  *EQ-5D Total = 1 - 0.081 - (the score of the each level) - 0.269 (if at least one of level 3 presents)
  EQ-5D total score could be 0.919 in maximum and -0.594 in minimum if case all index indicates the level 3. So, if EQ-5D total score closed by "1" means that the healthy condition and high quality of life.
Time Frame: Baseline and at 6 weeks
Population: In the PP set, the change in the quality of life (EQ-5D) total score from Visit 1 (Baseline) to Week 6 of the investigational product administration was analyzed.
Measure: Mean (Standard Deviation); unit: EQ-5D Total score
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Number analyzed (Participants) | 47 | 40
EQ-5D Total score | 0.09 (0.19) | 0.21 (0.22)

4. Secondary Outcome: Change From Baseline in Health-related Quality of Life Assessed by EuroQol Visual Analog Scale (EQ-5D VAS)
Description: The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' (score = 100) and 'Worst imaginable health state' (score = 0). Higher points were positive results and positive points of difference gap means improvement results.
Time Frame: Baseline and at 6weeks
Population: In the PP set, the change in the your today health score from Visit 1 (Baseline) to Week 6 of the investigational product administration was analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Number analyzed (Participants) | 47 | 40
scores on a scale | 14.33 (20.34) | 9.08 (19.63)

5. Secondary Outcome: Clinical Global Impression of Change(CGIC)
Description: The number of patients who choose the best opinion of overall satisfaction among Clinical Global Impression of Change Scale(CGIC) among 7 point scale. Missing data was imputed by LOCF. Scores measure from 1: Very much improved to 7:very much worse.
Time Frame: 6 weeks
Population: In the per protocol: Analyze the within-group change in the CGIC from Baseline (Week 0) to Week 6 of the investigational product administration by using a paired t-test, and analyze the between-group difference in the change of satisfaction by using a t-test.
Measure: Mean (Standard Deviation); unit: Scores on 1 to 7 point
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Number analyzed (Participants) | 47 | 40
Scores on 1 to 7 point | 2.28 (1.21) | 2.43 (1.01)

6. Secondary Outcome: Patient Global Impressions of Change(PGIC)
Description: In the PP set, Number of participants with categorical change in overall satisfaction.
  PGIC: a participant-rated instrument assessing change in participant's overall satisfaction from baseline, on a scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: 6 weeks
Population: Per protocol set: Analyze the within-group change in the PGIC from Baseline (Week 0) to Week 6 by using a paired t-test, and analyze the between-group difference in the change of satisfaction by using a t-test.
Measure: Mean (Standard Deviation); unit: Scores on 1 to 7point
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Number analyzed (Participants) | 47 | 40
Scores on 1 to 7point | 2.32 (1.22) | 2.45 (0.93)

ADVERSE EVENTS:
Time Frame: from baseline to 6 weeks
Groups:
- Buprenorphine: Patch
  buprenorphine: Dosage and administration: This one patch should be attached every 7 days.
  Safety was analyzed based on data for AEs, clinical laboratory tests, vital signs, and physical examination in the Safety set which consisted of 69 subjects who administered the study drug(buprenorphine) and had at least one time of safety assessment.
- Tramadol/Acetaminophen: Oral tablet
  tramadol/acetaminophen: Amount of drug ingredients
  : Acetaminophen 325 mg and Tramadol hydrochloride 37.5 mg in 1 tablet of this drug.
  Dosage and administration:
  Adjust dose depending on a patient's pain severity and treatment response. Starting at the initial dose of 2 tablets, usually administer 4 tablets per dose, twice daily. At a dosing interval of at least 12 hr, the daily dose should not exceed 8 tablets.
  Safety was analyzed based on data for AEs, clinical laboratory tests, vital signs, and physical examination in the Safety set which consisted of 65 subjects who administered the comparator(tramadol/acetaminophen) and had at least one time of safety assessment.
Arm/Group | Buprenorphine | Tramadol/Acetaminophen
Serious Adverse Events (participants affected / at risk) | 3/69 | 0/65
Other Adverse Events (participants affected / at risk) | 18/69 | 13/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (N=69) | Tramadol/Acetaminophen (N=65)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — This case was not related with study drug.
Post procedural infection (Infections and infestations) | 2 (2) | 0 (0) — These cases were not related with study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine (N=69) | Tramadol/Acetaminophen (N=65)
Constipation (Gastrointestinal disorders) | 4 (4) | 4 (4) — These cases were related with study drug & comparator.
Nausea (Gastrointestinal disorders) | 5 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 3 (3) | 0 (0)
Application site erythema (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Post procedural infection (Nervous system disorders) | 2 (2) | 0 (0)
Herpes zoster (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No